CLINICAL TRIAL: NCT00232570
Title: Quetiapine for the Treatment of Insomnia Associated With Alzheimer's Disease
Brief Title: Quetiapine for the Treatment of Insomnia in Alzheimer's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Vermont (Other)
Collaborators: AstraZeneca (Industry); National Center for Research Resources (NCRR) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 05-234
Record Dates: First submitted 2005-09-30; First posted 2005-10-04 (Estimated); Last update posted 2009-05-05 (Estimated); Status verified 2009-05

CONDITIONS: Alzheimer's Disease; Insomnia
Keywords: sleep disturbance; dementia
MeSH Terms: conditions — Alzheimer Disease; Sleep Initiation and Maintenance Disorders; Parasomnias; Dementia | interventions — Quetiapine Fumarate

STUDY DESIGN:
Who Masked: Participant

INTERVENTIONS:
Drug: quetiapine

SUMMARY:
The primary hypothesis is that quetiapine will improve sleep in persons with Alzheimer's Disease (AD), with higher doses producing greater total sleep time and sleep efficiency.

DETAILED DESCRIPTION:
Quetiapine is frequently used to treat psychosis in patients with Alzheimer's disease (AD) and other dementias. These patients commonly have sleep disturbances that include nighttime awakenings with confused, agitated behaviors. These awakenings impose a great challenge for caregivers, especially family caregivers whose own sleep is disrupted as a result of the patient's awakenings. Sleep disturbance can lead to nursing home placement3 and may add to cognitive impairment of patients.

There is no medication proven to be safe and effective in the treatment of sleep disorders in patients with dementia. Antipsychotic medications are often prescribed at bedtime in the hopes that they will aid sleep and reduce agitation and psychosis associated with these awakenings. Sleep disturbance is more common in AD patients with moderate to severe disease, and these patients are more likely to have psychosis and to be recruited from long-term care facilities. We recently conducted the only multicenter clinical trial of a drug for sleep disturbance in AD. The study, completed under the auspices of the NIA's Alzheimer's Disease Cooperative Study, investigated melatonin as a sedative-hypnotic agent for AD patients. We found melatonin to be of no benefit on objective measures, although there were positive trends in the data and a significant improvement on subjective measures (caregiver ratings of patients' sleep) in one of the melatonin groups relative to placebo. No other large trial in AD subjects has been reported in the literature for drugs with potential benefit for AD patients with sleep disturbances. There are several reasons why this population needs to be specifically studied. Patients with AD tend to have highly fragmented sleep, with many nocturnal awakenings. They have significant daytime sleepiness that might affect daytime cognitive function and behavior. These patients tend to be older, with sensitivity to drug side effects.

People with neurodegenerative diseases such as AD may respond differently to CNS-active medications. Finally, this population represents a large and growing cohort of patients that deserve individual study of their unique problems.

ELIGIBILITY:
Inclusion Criteria:

1. Age 55-90 years.
2. Diagnosis of possible or probable AD as defined by NINCDS-ADRD criteria.
3. Sleep disturbance defined by mean score of 3 on first six items of the SDI.
4. Family member able to provide surrogate informed consent.
5. Live-in caregiver able to monitor medication and serve as informant on questionnaires.
6. Caregiver who is fluent in English.
7. Be able to ingest oral tablets.
8. Be able to avoid caffeinated and alcoholic beverages during the study period.
9. A neuroimaging study at the time of initial diagnosis, or any time since that is consistent with AD and effectively rules out dementia related only to stroke, hydrocephalus or other neurological condition.

Exclusion Criteria:

1. Medical disorders that may account for sleep disturbance, especially delirium, Major Depressive Disorder (DSMIV) and severe or significant acute or chronic pain.
2. Have acute or unstable medical conditions including renal failure, abnormal liver function, cardiac arrhythmia, sitting blood pressure below 110/70 or above 140/100 or postural blood drop 20 mm Hg.
3. Symptoms suggesting other sleep disorders (e.g., periodic limb movement disorder, restless legs syndrome, obstructive sleep apnea syndrome), may be present but in the opinion of the PI, do not account for the primary symptoms of insomnia.
4. Sleep disturbance symptoms that suggest a parasomnia. Parasomnias may include behavioral manifestations of epileptiform activity or REM Behavior Disorder (RBD).
5. Previous treatment failure with quetiapine of AD-associated sleep disturbances, or intolerance of quetiapine in a previous treatment trial.
6. Concomitant treatment with another antipsychotic or sedative-hypnotic medication, including trazodone.
7. Evidence of a major mental disorder other than dementia, such as major depression or schizophrenia.
8. Stable doses (for 4 weeks prior to study entry) of antidepressant, antiepileptic mood stabilizer, or acetylcholinesterase inhibitor medication will be allowed, but initiation or recent changes in the dose of such medications will be prohibited.
9. Benzodiazepines within 2 weeks of study entry will not be allowed.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2005-11; Primary Completion 2009-12 (Estimated); Study Completion 2010-01 (Estimated)

PRIMARY OUTCOMES:
The primary objective is to determine whether quetiapine can increase total sleep time and reduce time awake in patients with AD and sleep disturbance.

SECONDARY OUTCOMES:
Dose-response relationship of quetiapine and sleep in AD patients?
Are there sleep architecture changes from quetiapine?
Do the primary sleep variables change relative to placebo at any weekly time or dose point?
Are caregivers, blind to treatment status, able to detect changes in sleep quality in the patients for quetiapine relative to placebo?
Does quetiapine used at single bedtime dosing for potential nighttime soporific effect have a measurable impact on neuropsychiatric symptoms other than insomnia?

CONTACTS AND LOCATIONS:
Overall Officials: Clifford Singer, M.D., Principal Investigator — University of Vermont
Locations (1):
- Fletcher Allen Health Care-Clinical Neuroscience Research Unit, Burlington, Vermont, United States